CLINICAL TRIAL: NCT00449709
Title: A Two-part, Open-label, Cross-over Study to Assess the Pharmacokinetics of GSK221149 Following Single Oral Doses of Various Modified Release Formulations and a Solution in Healthy Adult Subjects
Brief Title: A Study To Assess The Pharmacokinetics Of Different Modified Release Formulations Of GSK221149 In Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OTA106004
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Obstetric Labour, Premature; Premature Ejaculation
Keywords: Pre-term labor,; modified release formulation; pharmacokinetics,
MeSH Terms: conditions — Premature Birth; Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK221149

SUMMARY:
PreTerm Labor (prior to 37 weeks gestation) is the largest single cause of infant morbidity and mortality and is frequently associated with long-term disability. Oxytocin is a hormone produced by the body during labor. GSK221149 is an experimental drug that will be used to block the effects of oxytocin, and therefore pause or prevent contractions. In this study, the pharmacokinetics of various modified release formulations of GSK221149 will be investigated in healthy non-pregnant adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant female
* Between the ages of 18 and 50 years old.
* Females may be of child-bearing or non-child-bearing potential.
* Non-smokers
* BMI of between 19 and 30 kg/m2 (weight of greater than 110lbs).

Exclusion Criteria:

* History of smoking within past 6 months
* Regular alcohol consumption averaging 7 drinks or more per week
* Subject is positive for hepatitis C antibody, hepatitis B surface antigen, or HIV
* Use of prescription or non-prescription drugs within 14 days of study start

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Blood samples will be drawn and analyzed to assess how the body handles the drug over a 24 hour period during each study session. | over a 24 hour period during each study session.

SECONDARY OUTCOMES:
Safety and tolerability will be assessed by blood pressure, ECGs, and blood sampling over a 24 hour time period during each study session.. | over a 24 hour period during each study session.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States